CLINICAL TRIAL: NCT03992508
Title: The Effects of Compression and Massage Therapies in the Treatment of Breast Cancer-related Lymphoedema
Brief Title: Treatment of Breast Cancer-related Lymphoedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Engin Tastaban, Assistant Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/99
Record Dates: First submitted 2019-06-12; First posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- complex decongestive treatment (Other): In group 1, the patients were received standard complex decongestive therapy including skin care, manual lymphatic drainage, multi-layer compression bandaging and exercises. During the treatment, written and verbal information was given to the patients about skin care. Manual lymphatic drainage and compressive bandages were applied by a certified physical therapist. The patients received 30-minutes manual lymphatic drainage involving stationary circular, pumping, scooping, and rotary movements. Multi-layer compression bandaging was applied to the affected limb to promote the flow of excess interstitial fluid out of the extremity using a graded pressure for 22-23 hours in a day. The patients strictly followed a lymphoedema exercise program structured with breathing exercise, neck and shoulder range of motion, and stretching exercise to facilitating lymph resorption.
  Interventions: Procedure: complex decongestive therapy
- intermittent pneumatic compression (Experimental): In group 2, the patients received experimental intermittent pneumatic compression in addition to the standard complex decongestive therapy. The complex decongestive therapy procedure was the same as above, but additionally, 30 minutes of intermittent pneumatic compression was instituted using a pump (Pulse Press Multi 6 Pro; MJS Healthcare Ltd. UK) operating at 30-40 mmHg of pressure. All groups were given a total of 20 treatment sessions, including daily 5 times a week for 4 weeks.
  Interventions: Device: intermittent pneumatic compression; Procedure: complex decongestive therapy

INTERVENTIONS:
Device: intermittent pneumatic compression
  Arms: intermittent pneumatic compression
Procedure: complex decongestive therapy

SUMMARY:
To evaluate the role of intermittent pneumatic compression in the treatment of breast cancer-related lymphoedema.

DETAILED DESCRIPTION:
Patients with unilateral arm lymphoedema were enrolled and all were hospitalized. The participating patients were randomly divided into two groups.

Demographic features of the patients including age, body mass index [BMI = weight (kg) / height2 (m2)], duration of lymphoedema (months) and number of axillary lymph nodes removed were all recorded. The volume (V) of every part of the limb was calculated by the truncated cone formula according to circumferential measurements and the total volume is estimated by the sum of the increments. Circumference measurements were taken at 4-centimetre intervals along the arm from the level of the ulnar styloid to the shoulder with a flexible non-stretch tape measure. The volume between every two circumferential measurement levels was calculated using the following formula:

Volume = h (C2 + Cc + c2) / 12π In this formula, C is the first circumferential measurement (circumference of the top of the cone), c is the second circumferential measurement (circumference of the base of the cone) and h is the height from measurement C to c. Both the affected and non-affected limbs were evaluated by the same examiner. An Excel-based software program was used to convert these values into limb volumes in mL.

The severity of lymphoedema was characterized by the percentage excess volume (PEV) PEV = [(VLE - VH) / VH] x 100 where VLE denotes the volume of the lymphoedema arm and VH is that of the healthy arm. PEV is the preferred quantity for defining the severity of lymphoedema than the absolute difference volume. Also, this method minimizes the effects of BMI on the volume estimates. The efficacy of complex decongestive therapy, the response to the therapeutic intervention, was also quantified by the percentage reduction of excess volume (PREV) PREV = [(pre-treatment VLE - post-treatment VLE) / excess volume)] x 100. Other assessments of clinical origin were also conducted on the patients by physical therapists who were blind to the applied treatment and the timing of the data collection point. Pitting oedema was evaluated at multiple points on the forearm by pressing the thumb on the region to be investigated for a minute as hard as possible, as such test is considered as an indicator of the presence of excess free fluid accumulated in the superficial interstitial tissue spaces. The Stemmer's sign was performed as an inability to pinch the fold of skin at the base of the finger.

Clinical symptoms of pain (during activity, resting and night), heaviness and tightness in the affected arm were evaluated with Visual Analog Scale (VAS) with a 0-10 numerical rating scale. The patients' functional situation was assessed by the Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) outcome questionnaire which is a self-reported assessment tool for the measurement of physical function and symptoms in individuals with a musculoskeletal disorder of the upper limb. This instrument was also reported as a convenient, reliable, and valid patient-reported outcome measure to assess upper extremity disability in patients with breast cancer. The scores indicated the level of disability and severity, ranging from 0 (no disability) to 100 (most severe disability).

Grip strength was measured by using Jamar® hydraulic hand dynamometer (Sammons Preston, Bolingbrook, IL, USA). Both hands of the patient's grip strength were assessed by using the second level of resistant (3.75 cm) as the elbow is at 90º flexion, the forearm is in a neutral position. All measurements were performed bilaterally and three times. The average of the obtained values was recorded in kg. Beck Depression Inventory, a 21-item, self-administered inventory that measures clinical depression, was also administered to the patients. Scores ranged from 0 to 63, and higher scores were indicative of depression. The validity and reliability of the Beck Depression Inventory for the Turkish population have already been tested previously.

Kolmogorov-Smirnov test was used to test whether the data were normally distributed. All of the measured variables failed the normality test and thus median (25-75 percentiles) were given for nonparametric descriptive statistics. Wilcoxon T test was used for the intragroup comparison of the measurements between before and after the treatments. Mann-Whitney U-test was used for the intergroup comparison of the measurements after the treatments. Categorical variables were shown as number (%) and Chi-square tests were used for the comparison of categorical variables. P<0.05 was accepted as an indicator of the statistically significant difference.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer-related lymphoedema due to unilateral breast cancer
* more than 2 cm difference at the circumference measurements or >10% difference in volume between the two arms
* completed chemotherapy and radiotherapy

Exclusion Criteria:

* bilateral breast cancer
* primer lymphoedema
* undergone complex decongestive therapy or other interventions for lymphoedema within 12 months
* truncal and/or breast oedema
* continuing chemotherapy and/or radiotherapy
* active infection
* current metastases
* heart failure with arterial and/or venous occlusion
* elephantiasis
* impaired cognitive status
* received physiotherapy within last six months
* cervical or cranial originated upper extremity problems
* using any medications that affect the body fluid and electrolyte balance

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-08-17 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Change of excess arm volume from baseline | a month
  The volume of every part of the limb was calculated in liter by the truncated cone formula according to circumferential measurements.

SECONDARY OUTCOMES:
Change of arm pain, heaviness and tightness from baseline | a month
  The intensity of pain, heaviness and tightness were measured by visual analog scale (minimum score:0; maximum score:100)(higher values represent worse outcome)
Change of disability from baseline | a month
  The patients' functional situation was assessed by the Quick Disabilities of the Arm, Shoulder and Hand (Q-DASH) scale. The Q-DASH scores are ranging from 0 (no disability) to 100 (most severe disability).
Change of grip strength from baseline | a month
  The measurement of the grip strength in kg was performed by a hydraulic hand dynamometer.
Change of depression from baseline | a month
  The measurement of the depression was performed by the Beck Depression Inventory scoring.The scale is used to measure intensity and is a self-rating scale scored between 0 and 63. The cut-off point considered is 17. Higher scores reflect more severe depression.

IPD SHARING:
Plan to Share IPD: No